CLINICAL TRIAL: NCT03469843
Title: Characterization of the Cardiac Reinnervation of Patients With Transposition of the Great Arteries Long After Repair With the Arterial Switch Operation. Correlation With Electrocardiographic and Exercise Test Parameters
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AMI)126/2015
Record Dates: First submitted 2018-02-20; First posted 2018-03-19 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Congenital Heart Disease; Congenital Heart Defect; Transposition of the Great Arteries
Keywords: Congenital Heart Disease; Cardiac denervation; 123I-metaiodobenzylguanidine; Arterial switch operation
MeSH Terms: conditions — Heart Defects, Congenital; Transposition of Great Vessels | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: patients with transposition of the great arteries long after repair with the arterial switch operation
  Interventions: Other: Non intervention

INTERVENTIONS:
Other: Non intervention — patients without intervention
  Other Names: patients without intervention

SUMMARY:
Cardiac denervation is inherent to the arterial switch (ASO) technique for the repair of transposition of the great arteries (TGA) and the long term reinnervation process has not been studied. We sought to describe the reinnervation status of adult patients long after the ASO, to identify areas of myocardial perfusion/innervation mismatch and to assess the relation of innervation status and exercise capacity.

DETAILED DESCRIPTION:
Cardiac denervation is inherent to the arterial switch (ASO) technique for the repair of transposition of the great arteries (TGA) and the long term reinnervation process has not been studied. We sought to describe the reinnervation status of adult patients long after the ASO, to identify areas of myocardial perfusion/innervation mismatch and to assess the relation of innervation status and exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with transposition of the great arteries repaired with the arterial switch.
* Patients aged of more than 18 years-old.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Denial of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged of more than 18 years-old with transposition of the great arteries repaired with the arterial switch
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Myocardial innervation pattern on 123I-mlBG SPECT. | 1 day
  To describe the myocardial reinnervation pattern of a cohort of patients with TGA long after ASO using cardiac nuclear imaging.

SECONDARY OUTCOMES:
Myocardial perfusion defects on cardiac nuclear imaging. | 1 day
  To identify myocardial perfusion defects using cardiac nuclear imaging.
Myocardial innervation perfusion mismatch defects on cardiac nuclear imaging. | 1 day
  To identify myocardial innervations/perfusion mismatch using cardiac nuclear imaging.
Treadmill exercise test. | 1 day
  To determine exercise capacity (METs and double product) and chronotropic response (Maximal heart rate and heart rate increase pattern). Correlate with myocardial reinnervation pattern and sinus node reinnervation.
  To determine exercise induced ischeamic ST segment changes. Correlate with myocardial perfusion defects and innervation-perfusion mismatch.
24 hours ECG Holter monitoring . | 1 day
  To determine sinus node innervation through heart rate variability (HRV) which will be assessed by time domain variables (the standard deviation of normal RR intervals (SDNN) and the square root of the mean of the squared differences between adjacent normal RR intervals (r-MSSD)) and frequency domain variables (variance of all R-R intervals - total power (TP); power in the very low frequency range - very low frequency (VLF, 0.003-0.04 Hz); power in the low frequency range-low frequency (LF, 0.04-0.15Hz); low frequency power in normalized units-normalized low frequency; power in the high frequency range-high frequency (HF, 0.15-0.40 Hz); and high frequency power in normalized units-normalized high frequency and the ratio of low frequency to high frequency (LF/HF)).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dos Subirà, PhD MD, Principal Investigator — Hospital Universitari Vall d'hebron Barcelona, Spain
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tobler D, Williams WG, Jegatheeswaran A, Van Arsdell GS, McCrindle BW, Greutmann M, Oechslin EN, Silversides CK. Cardiac outcomes in young adult survivors of the arterial switch operation for transposition of the great arteries. J Am Coll Cardiol. 2010 Jun 29;56(1):58-64. doi: 10.1016/j.jacc.2010.03.031. PMID 20620718
- [Result] Khairy P, Clair M, Fernandes SM, Blume ED, Powell AJ, Newburger JW, Landzberg MJ, Mayer JE Jr. Cardiovascular outcomes after the arterial switch operation for D-transposition of the great arteries. Circulation. 2013 Jan 22;127(3):331-9. doi: 10.1161/CIRCULATIONAHA.112.135046. Epub 2012 Dec 12. PMID 23239839
- [Result] Kondo C, Nakazawa M, Momma K, Kusakabe K. Sympathetic denervation and reinnervation after arterial switch operation for complete transposition. Circulation. 1998 Jun 23;97(24):2414-9. doi: 10.1161/01.cir.97.24.2414. PMID 9641693
- [Result] Grupper A, Gewirtz H, Kushwaha S. Reinnervation post-heart transplantation. Eur Heart J. 2018 May 21;39(20):1799-1806. doi: 10.1093/eurheartj/ehw604. PMID 28087606